CLINICAL TRIAL: NCT04782102
Title: SOPHIE: a Randomised Controlled Trial to Investigate the Efficacy of Online-intervention for Prevention and Treatment of Social Anxiety in Adolescents
Brief Title: SOPHIE: Online-intervention for Prevention and Treatment of Social Anxiety in Adolescents
Acronym: SOPHIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-02501
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Social Anxiety; Social Anxiety Disorder
Keywords: Prevention; Intervention; Adolescents; Youths; Online-Intervention; Internet-Intervention
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOPHIE Intervention (Experimental): SOPHIE is an online-intervention aiming to reduce social anxiety in adolescents. SOPHIE has 8 modules, one module per week, which lasts about 60 minutes. SOPHIE includes elements of evidence-based psychotherapeutic interventions to reduce social anxiety and of an existing online-intervention for adults with social anxiety adopted to the needs of adolescents. The intervention consists of psychoeducation (how social anxieties arise), application examples (e.g. setting up a personal anxiety cycle or anxiety pyramid, imagination exercise: journey to a safe place), and contains weekly tasks for which regular repetition in everyday life is important (e.g. progressive muscle relaxation, observing anxiety in everyday life, exposures in various situations). At the end of each module, a short quiz allows participants to recall and consolidate what they have learned. The content is presented in video inputs, short explanatory texts, application tasks and quizzes.
  Interventions: Behavioral: SOPHIE Intervention
- Care-as-usual (No Intervention): Care-As-Usual: all other kinds of interventions are allowed and will be recorded using the Client Sociodemographic and Service Receipt Inventory (Chisholm et al., 2000; Roick et al., 2001)

INTERVENTIONS:
Behavioral: SOPHIE Intervention — SOPHIE is an online-intervention aiming to reduce social anxiety in adolescents. SOPHIE has 8 modules, one module per week, which lasts about 60 minutes. SOPHIE includes elements of evidence-based psychotherapeutic interventions to reduce social anxiety and of an existing online-intervention for adults with social anxiety adopted to the needs of adolescents. The intervention consists of psychoeducation (how social anxieties arise), application examples (e.g. setting up a personal anxiety cycle or anxiety pyramid, imagination exercise: journey to a safe place), and contains weekly tasks for which regular repetition in everyday life is important (e.g. progressive muscle relaxation, observing anxiety in everyday life, exposures in various situations). At the end of each module, a short quiz allows participants to recall and consolidate what they have learned. The content is presented in video inputs, short explanatory texts, application tasks and quizzes.
  Arms: SOPHIE Intervention

SUMMARY:
This study's aim is to investigate the efficacy of the online-intervention SOPHIE. SOPHIE is an online-intervention for adolescents with social anxiety. In Switzerland, Germany, Austria and Liechtenstein, about one in 15 adolescents suffers from social anxiety. The SOPHIE intervention aims to help these adolescents to better understand and cope with their social anxiety symptoms and to feel more comfortable in social situations. The investigators intend to include 248 adolescents in the study. Stratified by subclinical and clinical level of social anxiety, participants will be randomly assigned to the SOPHIE group or the control group receiving care-as-usual. Both groups will complete online questionnaires and will be interviewed via telephone several times during the study. This allows to compare the two groups regarding their efficacy of the SOPHIE programme in terms of changes in social anxiety over time.

ELIGIBILITY:
Inclusion Criteria:

* Age between 11;00 (11 years and 0 months) and 17;11 (17 years and 11 months)
* Good written and spoken German language skills
* Access to an Internet connection and a device to use the intervention (tablet, smartphone, PC) and to collect the EMA data (smartphone)
* Subclinical values on the SPIN (value: 16-23; Loscalzo et al., 2018) or criteria for social anxiety disorder according to Kinder-DIPS (Schneider et al., 2017)
* Written consent of the adolescent (if at least 14 years old) or the parents or guardian (if adolescent under 14 years old) and assent of adolescent under 14 years old

Exclusion Criteria:

* Known diagnosis of autism spectrum disorder
* Current suicidal ideation (collected via PHQ-A Item 9)
* Lack of knowledge of the German language in spoken and written form
* Past diagnosis of social anxiety according to the DSM-5 criteria assessed by the Kinder-DIPS (Schneider et al., 2017) in participants with current subclinical anxiety

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in social anxiety assessed by the Social Phobia Inventory (SPIN; Connor et al., German Version: Sosic et al., 2008) | Baseline assessment compared to assessment at post-intervention (2 months after baseline)
  Measure of social anxiety, total score ranging from 0 - 68 (representing the sum of each of the 17 individual items). Lower scores represent less social anxiety and a more favourable outcome.

SECONDARY OUTCOMES:
Current and past mental disorder assessed by the structured diagnostic interview for mental disorders of childhood and adolescence (Kinder-DIPS; Schneider et al., 2017) | Assessed at baseline, at post-intervention (2 months after baseline) and follow-up (5 months after intervention);
  At Baseline, the entire Kinder-DIPS will be assessed. At post and follow-up, only the sections for social anxiety and comorbid diagnoses met at baseline are assessed.
Change in global functioning assessed by the GF Social (Cornblatt et al., 2007) | Assessed at baseline, at post-intervention (2 months after baseline) and follow-up (5 months after intervention)
  Structured interview assessing the level of functioning in social areas of life (friends & family) ranging from 1 to 10, higher scores indicate a better level of functioning
Change in global functioning assessed by the GF Role Scale (Cornblatt et al., 2007) | Assessed at baseline, at post-intervention (2 months after baseline) and follow-up (5 months after intervention)
  Structured interview assessing the level of functioning in school / work ranging from 1 to 10, higher scores indicate a better level of functioning
Utilisation of help assessed by the Client Sociodemographic and Service Receipt Inventory (CSSRI-EU; Chisholm et al., 2000; Roick et al., 2001) | Assessed at post-intervention (2 months after baseline) and follow-up (5 months after baseline)
  Structured interview assessing the additional use of psychological, medical and other formal and informal services and sources of help (e.g. at school, friends)
Change of fear of negative evaluation and avoidance assessed by the Social Anxiety Scale for Adolescents (SAS-A; La Greca & Lopez,1998) | Assessed at baseline, at mid-treatment (1 month after baseline), at post-intervention (2 months after baseline), and at follow-up (5 months after baseline)
  Total score ranging from 18 - 90 (representing the sum of each of the 18 individual items). Lower scores represent less fear of negative evaluation and avoidance and a more favourable outcome.
Change of generalized anxiety symptoms assessed by the Generalized Anxiety Disorder 7 (GAD-7; Löwe et al., 2008) questionnaire | Assessed at baseline, at mid-treatment (1 month after baseline), at post-intervention (2 months after baseline), and at follow-up (5 months after baseline)
  Total score ranging from 7 - 35 (representing the sum of each of the 7 individual items). Lower scores represent less anxiety and a more favourable outcome.
Change in depressive symptoms assessed by the Patient Health Questionnaire-9 for Adolescents (PHQ-A; Johnson et al., 2002) | Assessed at baseline, at mid-treatment (1 month after baseline), at post-intervention (2 months after baseline), and at follow-up (5 months after baseline)
  Total score ranging from 0 - 27 (representing the sum of each of the 9 individual items). Lower scores represent less depressive symptoms and a more favourable outcome.
Change in health-related quality of life assessed by the KIDSCREEN-10 (Ravens-Sieberer et al., 2010) | Assessed at baseline, at mid-treatment (1 month after baseline), at post-intervention (2 months after baseline), and at follow-up (5 months after baseline)
  Total score ranging from 11 - 55 (representing the sum of each of the 11 individual items). Higher scores represent a higher quality of life and a more favourable outcome.
Change in self-esteem assessed by the Rosenberg Self-Esteem Scale (RSES; Rosenberg, 1965) | Assessed at baseline, at mid-treatment (1 month after baseline), at post-intervention (2 months after baseline), and at follow-up (5 months after baseline)
  Total score ranging from 0 - 30 (representing the sum of each of the 10 individual items). Higher scores represent a higher self-esteem and a more favourable outcome.
Change in social anxiety assessed by the Social Phobia Inventory (SPIN; Connor et al., German Version: Sosic et al., 2008) | Assessed at baseline, at mid-treatment (1 month after baseline), at post-intervention (2 months after baseline), and at follow-up (5 months after baseline)
  Measure of social anxiety, total score ranging from 0 - 68 (representing the sum of each of the 17 individual items). Lower scores represent less social anxiety and a more favourable outcome.

OTHER OUTCOMES:
Adherence to the Online-Intervention | During the eight-week online-intervention
  Assessed within the online-intervention. Indicator of adherence: time spent in program.
Adherence to the Online-Intervention | During the eight-week online-intervention
  Assessed within the online-intervention. Indicator of adherence: number of clicks.
Adherence to the Online-Intervention | During the eight-week online-intervention
  Assessed within the online-intervention. Indicator of adherence: number of modules completed.
Adherence to the Online-Intervention | During the eight-week online-intervention
  Assessed within the online-intervention. Indicator of adherence: number of exercises completed.
Negative effects of the online-intervention | Assessed at post-intervention (2 months after baseline)
  Assessed with the Inventar zur Erfassung Negativer Effekte in der Psychotherapie für Kinder (Kinder-INEP; Bieda et al., 2018). Total score ranging from -3 - 38 (representing the sum of each of the 15 individual items). Higher scores represent more negative effects of the online-intervention and a less favourable outcome.
Satisfaction with the online-intervention assessed by the Zufriedenheit mit der Intervention (ZUF-8; Schmidt et al., 1989) questionnaire | Assessed at post-intervention (2 months after baseline)
  Total score ranging from 8 - 32 (representing the sum of each of the 8 individual items). Higher scores represent more satisfaction and a more favourable outcome.
Therapeutic alliance assessed by the Working Alliance Inventory for Guided Internet Interventions (WAI-I; Gómez Penedo et al., 2020) | Assessed 2, 4, 6, and 8 weeks after baseline (during the online-intervention every two weeks)
  Total score ranging from 12 - 60 (representing the sum of each of the 12 individual items). Higher scores represent a higher working alliance and a more favourable outcome.
Motivation of adolescent for the online-intervention assessed with the Motivation for Youth's Treatment Scale (MYTS; Breda & Riemer, 2012) youth version | Assessed at baseline and every two week during the eight week online-intervention (after 2, 4, 6, and 8 weeks)
  Total score ranging from 8 - 40 (representing the sum of each of the 8 individual items). Higher scores represent more motivation and a more favourable outcome.
Motivation of parent / guardian for the online-intervention assessed with the Motivation for Youth's Treatment Scale (MYTS; Breda & Riemer, 2012) parent version | Baseline, mid-intervention(after 1 Month), and at post-intervention (after 2 months)
  Total score ranging from 8 - 40 (representing the sum of each of the 8 individual items). Higher scores represent more motivation and a more favourable outcome.
Adolescents' expectation of the online-intervention assessed with the Credibility/Expectancies Questionnaire (CEQ; Devilly & Borkovec, 2000) youth version | Assessed at baseline
  Total score ranging from 4 - 36 (representing the sum of each of the 4 individual items) and two items indicating percents from 0-100. Higher scores represent higher expectations of the online-intervention.
Parents' / Guardians' expectation of the online-intervention assessed with the Credibility/Expectancies Questionnaire (CEQ; Devilly & Borkovec, 2000) parent version | Assessed at baseline
  Total score ranging from 4 - 36 (representing the sum of each of the 4 individual items) and two items indicating percents from 0-100. Higher scores represent higher expectations of the online-intervention.
Ecological Momentary Assessment (EMA) | 3 times a day during the eight week online-intervention, and three times a day for the two succeeding weeks after the follow-up assessment (5 months after baseline).
  The Ecological Momentary Assessment consists of 20 short questions asking about the momentary social context, the momentary affect (Positive and negative affective schedule for children; PANAS-C; Ebesutani et al., 2012) and factors maintaining social anxiety (derived from the Social phobia weekly summary scale; SPWSS; Clark et al., 2003).
Change in parents' / guardians' assessment of their children's social anxieties assessed by the Elternfragebogen zu sozialen Ängsten im Kindes- und Jugendalter (ESAK, van Gemmeren et al., 2008) | Assessed at baseline, at mid-treatment (1 month after baseline), at post-intervention (2 months after baseline), and at follow-up (5 months after baseline)
  Total score ranging from 18 - 72 (representing the sum of each of the 18 individual items). Lower scores represent less social anxiety and a more favorable outcome.
Interview with adolescents in the intervention group on satisfaction with the online intervention | Assessed at post-intervention (2 months after randomization)
  Qualitative Interview

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie J Schmidt, Prof. Dr., Principal Investigator — University of Bern; Thomas Berger, Prof. Dr., Study Chair — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Walder N, Berger T, Schmidt SJ. Prevention and Treatment of Social Anxiety Disorder in Adolescents: Protocol for a Randomized Controlled Trial of the Online Guided Self-Help Intervention SOPHIE. JMIR Res Protoc. 2023 Jun 21;12:e44346. doi: 10.2196/44346. PMID 37342086
- See also: Website of the online-intervention SOPHIE — https://selfhelp.psy.unibe.ch/sophie/homepage